CLINICAL TRIAL: NCT03098147
Title: The Influence of Benign Prostatic Hyperplasia on Bladder Function: A Multi-centre, Prospective and Case-control Study
Brief Title: The Influence of Benign Prostatic Hyperplasia on Bladder Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangfu Zhou (Other)
Responsible Party: Sponsor-Investigator, Xiangfu Zhou, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: Xzhou
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lower urinary tract symptoms(LUTS) are the main symptoms of benign prostatic hyperplasia(BPH), a benign but progressive disease which can advance to be with overactive bladder(OAB) symptoms. Moreover, LUTS and OAB symptoms can badly influence patients' especially the elderly's quality of life. Therefore, it appears to be urge to carry out researches on the functional impairment of bladder along with the advance of BPH. Besides, the management aimed at improving the LUTS and OAB symptoms come to be the key one among the management of BPH. For a long period, medication and surgery sustain to be the two most common therapies for BPH patients. Both patients and urologists prefer pharmacotherapeutics to surgery，which contributes to the rising number of BPH patients companied with OAB symptoms and storing symptoms complaint post-surgery. In fact, investigators usually find bladder impairment macroscopically in the BPH surgery: mild may be the trabeculation, worse can be the cabin, and severe may be the diverticula. Furthermore, it's not uncommon that patients with a long BPH history continually suffer from dysuria after surgery due to the detrusor muscle weakness. Consequently, investigators need to catch a moment when investigators should operate on such a patient in order to harvest a satisfying outcome. And perhaps the moment should be ahead of the existing guideline suggests. Thus, for understanding the influence of BPH on bladder function, investigators plan to conduct a prospective, case-control study recruiting in-patients with different degree of obstruction. Our team wish that such a clinical trail could provide valuable evidence for us to find out relatively better operating timing and serial indications. For the purpose of improving the quality of life and prolong life-span, investigators design the study above to maximum the operating outcome and minimize the bladder dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent.
2. The BPH in-patients who take 'dysuria' as the main self-reported symptom and meet the following conditions, 1) Maximal urinary flow rate less than 20 ml per second, 2) Volume of prostate more than 20ml measured by transrectal ultrasound 3) PSA ranges from 0 to 10ng/ml 4) IPSS>1

Exclusion Criteria:

1. The lower urinary tract obstruction caused not by BPH
2. Had a history of prostate cancer, surgery for benign prostatic hyperplasia or neurogenic bladder.
3. using medications known to affect urination or had a severe concomitant disease

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BPH in-patients from more than ten hospitals in southern China
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
IPSS | 1 year
  International Prostate Symptom Score

SECONDARY OUTCOMES:
Qmax | 1 year
  Maximum flow rate
RUV | 1 year
  residual urine volume
OABSS | 1 year
  Overactive Bladder Symptom Score

CONTACTS AND LOCATIONS:
Overall Officials: Xiangfu Zhou, Professor, Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No